CLINICAL TRIAL: NCT06884774
Title: Hemorrhoidectomy With or Without Lateral Internal Sphincterotomy in Management of Patients With Hemorrhoids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mohamed Salah, Lecturer of General Surgery, Faculty of Medicine, Minia University, Minia, Egypt., Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1230/08/2024
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Lateral Internal Sphincterotomy; Hemorrhoidectomy; Hemorrhoids
MeSH Terms: conditions — Hemorrhoids | interventions — Hemorrhoidectomy; Lateral Internal Sphincterotomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lateral internal sphincterotomy group (Experimental): Patients undergoing Hemorrhoidectomy with lateral internal sphincterotomy.
  Interventions: Procedure: Hemorrhoidectomy with lateral internal sphincterotomy
- Control group (Active Comparator): Patients undergoing Hemorrhoidectomy without lateral internal sphincterotomy.
  Interventions: Procedure: Hemorrhoidectomy

INTERVENTIONS:
Procedure: Hemorrhoidectomy with lateral internal sphincterotomy — Patients undergoing Hemorrhoidectomy with lateral internal sphincterotomy.
  Arms: Lateral internal sphincterotomy group
Procedure: Hemorrhoidectomy — Patients undergoing Hemorrhoidectomy without lateral internal sphincterotomy.
  Arms: Control group

SUMMARY:
This study aims to compare the lateral internal sphincterotomy versus no lateral internal sphincterotomy during hemorrhoidectomy in the management of patients with hemorrhoids.

DETAILED DESCRIPTION:
Hemorrhoidectomy is associated with postoperative pain, and no single surgical technique has been proven to reduce the pain significantly.

However, there are many drawbacks to such techniques, such as postoperative pain and constipation. The cause of this postoperative pain is multifactorial. Spasm of the internal anal sphincter (IAS) is one of the factors which is exposed and impinged after EH. Therefore, Lateral internal sphincterotomy (LIS) is a widely used adjunct treatment after EH, which can abolish spasms of the IAS and subsequently relieve postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years old.
* Both sexes.
* All patients indicated for surgical Hemorrhoidectomy (2nd, 3rd, and 4th degree piles).

Exclusion Criteria:

* Patients with 1st degree piles.
* Patients with piles plus fissure.
* Age above 70 years old
* Unfit for surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Anal pain score | 4 weeks postoperatively
  The pain was measured by visual analog scoring (VAS) described as : 0-no pain, at score 1 to 3- mild pain, score 4 to 6-moderate pain, at score 7 to 10- severe pain. Post-operative pain was observed on subsequent visits after 48 hours, one week and 4 weeks postoperatively.

SECONDARY OUTCOMES:
Degree of incontinence | 48 hours postoperatively.
  Incontinence was assessed by Wexner's incontinence score for solid, liquid, and gas until 48 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.